CLINICAL TRIAL: NCT06639217
Title: Comprehensive Nursing Care Protocol for Women With Pelvic Organ Prolapse and Urinary Incontinence: A Global Perspective
Acronym: Nurse Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Women Pelvic Organ Prolapse
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: women prolapse -Care Protocol
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a comprehensive nursing care protocol (Experimental): a comprehensive nursing care protocol provided for nurses who provide direct care for women with pelvic organ prolapse and urinary incontinence on their knowledge and practices as well as its impact on the women quality of life
  Interventions: Other: a comprehensive nursing care protocol

INTERVENTIONS:
Other: a comprehensive nursing care protocol — a comprehensive nursing care protocol provided for nurses who provide direct care for women with pelvic organ prolapse and urinary incontinence on their knowledge and practices as well as its impact on the women quality of life

SUMMARY:
Pelvic organ prolapse is the descent of pelvic structures into the vagina due to ligament or muscular weakness. Pelvic organ prolapse (POP) is subcategorized according to the compartment of descent. Cystocele characterizes anterior wall herniation, rectocele refers to the posterior vaginal wall descent, and vaginal vault prolapse characterizes the descent of the uterus, cervix, or apex of the vagina. They can occur either singly or in combination

DETAILED DESCRIPTION:
this study aimed to investigate the effectiveness of a comprehensive nursing care protocol provided for nurses who provide direct care for women with pelvic organ prolapse and urinary incontinence in gynecological in patients departments, Mansoura University Hospital, Mansoura University on their knowledge and practices as well as its impact on the women quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All available nurses assigned for bed side care in the previous study settings and fulfilled the following inclusion criteria:

  * Age 20≥ 60 years
  * Willing to participate in the study
  * Both sex

Exclusion Criteria:

* nurses did not assign for bed side care in the previous study settings and not fulfill the inclusion criteria

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-08-02 (Actual); Study Completion 2025-08-03 (Actual)

PRIMARY OUTCOMES:
Nurses knowledge structured interview | 3 months
  two main parts.
  Part I: Lifestyle interventions:
  This part will be including items related to weight loss, reducing exacerbating activities (e.g. heavy lifting, coughing) and treating constipation, pelvic floor muscle exercises etc.)
  Part II: pessaries intervention:
  This part will be including items related to indication of pessaries use, pessary maintenance and follow-up, complications, various types of pessaries, etc.) The scoring system. This tool will be scored on 2 point Likert scale . The researcher will give (1) point for each correct answer and (0) point for each incorrect answer, or don't know.
  Total knowledge score will be summed, transferred to percent and categorized as follows:
  * poor (<50% of the total score)
  * fair (50-≤80% of the total score)
  * good (≥80
Nurses Observational Practices Checklist | 3 months
  This tool will be scored on 4 point Likert scale for each item as follows:
  * Done correctly and completely (3)
  * Done but incompletely (2).
  * Done incorrectly (1).
  * Not done (0). The total score for nurses' practices was classified as the following;
    * A score of more than 75% was considered "Satisfactory nursing practices".
    * A score of less than 75% was considered "Unsatisfactory nursing practices".

CONTACTS AND LOCATIONS:
Locations (1):
- Basma, Al Mansurah, Al Dakahlia,, Egypt